CLINICAL TRIAL: NCT01600729
Title: Reliability of the Facial Wrinkle Scale in Japanese Subjects
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-119
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Facial Rhytides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants with facial lines. There was no intervention in this study.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — No intervention.

SUMMARY:
This study will evaluate the inter-rater and intra-rater reliability of the Facial Wrinkle Scale with Asian Photonumeric Guide (FWS-A) in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to assess facial lines in a mirror
* Removal of facial jewelry and makeup for study visit

Exclusion Criteria:

* Infection or skin disorder affecting the face
* Planned use of botulinum toxin of any serotype between Screening and Day 1
* Planned facial cosmetic procedure between Screening and Day 1
* Planned excessive/prolonged sun exposure between Screening and Day 1

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with facial lines
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 66
Completed | 65
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 66
Age Continuous [Median (Full Range); unit: Years] | 52.5 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability of Assessment of Facial Lines Using the 4-Point Facial Wrinkle Scale (FWS-A)
Description: Inter-rater (among raters) agreement of the FWS-A scores (0= none; 1= mild; 2= moderate; 3= severe) was evaluated by Kappa statistics. Kappa statistics were calculated for each of 7 raters who evaluated 66 participant's severity of facial lines in 4 areas (Glabellar Lines, Forehead Lines, Crow's Feet Lines on the Left side of the face and Crow's Feet Lines on the Right side of the face) at rest and maximum expression using the FWS-A scale. The overall inter-rater agreement for Kappa statistics for all raters combined was estimated by pooling Kappa statistics for each rater using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was predefined as: ≤ 0= poor, 0.00-0.20= slight, 0.21-0.40= fair, 0.41-0.60= moderate, 0.61-0.80= substantial and 0.81-1.00= almost perfect. The 95% confidence interval for Kappa statistics was provided.
Time Frame: Day 1
Population: Reliability population included all enrolled participants with at least 1 assessment by at least 1 live rater performed on day 1.
Measure: Mean (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 66
Kappa statistics
  Forehead Lines at Rest | 0.653 [0.621 to 0.684]
  Glabellar Lines at Rest | 0.637 [0.607 to 0.668]
  Crow's Feet Left Side at Rest | 0.647 [0.616 to 0.678]
  Crow's Feet Right Side at Rest | 0.654 [0.623 to 0.685]
  Forehead Lines at Maximum Brow Elevation | 0.527 [0.495 to 0.560]
  Glabellar Lines at Maximum Frown | 0.507 [0.473 to 0.540]
  Crow's Feet Left Side at Maximum Smile | 0.641 [0.610 to 0.671]
  Crow's Feet Right Side at Maximum Smile | 0.622 [0.592 to 0.653]

2. Primary Outcome: Intra-rater Reliability of Assessment of Facial Lines Using the 4-Point Facial Wrinkle Scale (FWS-A)
Description: Intra-rater (within raters) agreement of the FWS-A scores (0=none; 1=mild; 2=moderate; 3=severe) was evaluated by weighted Kappa statistics (WKS). WKS were calculated for each of 7 raters who evaluated 65 participant's severity of facial lines in 4 areas (Glabellar Lines, Forehead Lines, Crow's Feet Lines on the Left side of the face and Crow's Feet Lines on the Right side of the face) at rest and maximum expression using the FWS-A scale at 2 different time-points on Day 1. The overall intra-rater agreement for WKS for all raters combined was estimated by pooling WKS for each rater using a chi-square statistic. The degree of agreement of the point estimates of WKS was interpreted according to the reference range scale that was predefined as: ≤0=poor, 0.00-0.20=slight, 0.21-0.40=fair, 0.41-0.60=moderate, 0.61-0.80=substantial and 0.81-1.00=almost perfect. The 95% confidence interval for WKS was provided.
Time Frame: Day 1
Population: Participants from the Reliability population (all enrolled participants with at least 1 assessment by at least 1 live rater performed on day 1) who had 2 assessments on Day 1 available for analysis.
Measure: Mean (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 65
Kappa statistics
  Forehead Lines at Rest | 0.886 [0.858 to 0.914]
  Glabellar Lines at Rest | 0.861 [0.832 to 0.890]
  Crow's Feet Left Side at Rest | 0.841 [0.809 to 0.872]
  Crow's Feet Right Side at Rest | 0.838 [0.806 to 0.869]
  Forehead Lines at Maximum Brow Elevation | 0.810 [0.775 to 0.846]
  Glabellar Lines at Maximum Frown | 0.770 [0.731 to 0.808]
  Crow's Feet Left Side at Maximum Smile | 0.836 [0.804 to 0.867]
  Crow's Feet Right Side at Maximum Smile | 0.832 [0.800 to 0.864]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.